CLINICAL TRIAL: NCT04888845
Title: Refinement of Suicide Risk Management Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Monika Lohani, Assistant Professor, University of Utah
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00135355
Record Dates: First submitted 2021-04-29; First posted 2021-05-17 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Structured Interview; Narrative Assessment; Safety Plan; Crisis Response Plan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Structured interview and Safety Plan (Active Comparator): In the structured interview approach, clinicians ask a series of predetermined questions and/or assess a specified set of risk and protective factors, typically using a checklist-based approach. The safety plan is a written, prioritized list of coping strategies and resources for reducing suicide risk.
  Interventions: Behavioral: Safety Plan; Behavioral: Structured interview
- Structured interview and Crisis Response Plan (Active Comparator): In the structured interview approach, clinicians ask a series of predetermined questions and/or assess a specified set of risk and protective factors, typically using a checklist-based approach. Crisis response planning intervention teaches a range of coping strategies and provides support that can reduce suicide attempts and ideation.
  Interventions: Behavioral: Crisis Response Plan; Behavioral: Structured interview
- Narrative assessment and Safety Plan (Active Comparator): In the narrative assessment approach, clinicians ask patients to "tell the story" of their suicidal crisis. The safety plan is a written, prioritized list of coping strategies and resources for reducing suicide risk.
  Interventions: Behavioral: Safety Plan; Behavioral: Narrative Assessment
- Narrative assessment and Crisis Response Plan (Active Comparator): In the narrative assessment approach, clinicians ask patients to "tell the story" of their suicidal crisis. Crisis response planning intervention teaches a range of coping strategies and provides support that can reduce suicide attempts and ideation.
  Interventions: Behavioral: Crisis Response Plan; Behavioral: Narrative Assessment

INTERVENTIONS:
Behavioral: Safety Plan — The safety plan is a written, prioritized list of coping strategies and resources for reducing suicide risk.
  Arms: Narrative assessment and Safety Plan; Structured interview and Safety Plan
Behavioral: Crisis Response Plan — Crisis response planning intervention teaches a range of coping strategies and provides support that can reduce suicide attempts and ideation.
  Arms: Narrative assessment and Crisis Response Plan; Structured interview and Crisis Response Plan
Behavioral: Structured interview — In the structured interview approach, clinicians ask a series of predetermined questions and/or assess a specified set of risk and protective factors, typically using a checklist-based approach.
  Arms: Structured interview and Crisis Response Plan; Structured interview and Safety Plan
Behavioral: Narrative Assessment — In the narrative assessment approach, clinicians ask patients to "tell the story" of their suicidal crisis.
  Arms: Narrative assessment and Crisis Response Plan; Narrative assessment and Safety Plan

SUMMARY:
Participants will be randomly assigned to 1 of the 4 interventions using a sequential stratified randomization procedure. We will use sex (M, F) and history of suicide attempts (never, 1, and multiple) as our randomization strata. Participants will be assessed before and after the intervention to study the potential effects of each approach on suicide-related clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of suicide Ideation
* History of suicide attempts

Exclusion Criteria:

* Geographic location outside the U.S.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in suicide relevant thoughts and behaviors after the intervention (Self Injurious Thoughts and Behaviors questionnaire) | During an average of 2-weeks pre-intervention, 2-weeks post-intervention, 1 month follow-up after intervention
  Items from the Self Injurious Thoughts and Behaviors questionnaire (Fox et al., 2020) will be used to assess suicide relevant thoughts and behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Monika Lohani, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - The Ohio State, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lohani M, Baker JC, Elsey JS, Dutton S, Findley SP, Langenecker SA, Do AS, Bryan CJ. Suicide prevention via telemental health services: insights from a randomized control trial of crisis response plan and self-guided safety planning approaches. BMC Health Serv Res. 2024 Nov 12;24(1):1389. doi: 10.1186/s12913-024-11739-w. PMID 39533271